CLINICAL TRIAL: NCT05807061
Title: Reducing Children's Racial Biases Via a Parent-Led Intervention
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2020-1026; 1R01HD106970-01A1 (NIH); Psychology (Other: UW Madison)
Record Dates: First submitted 2023-03-29; First posted 2023-04-10 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Racial Bias
MeSH Terms: conditions — Racism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EmBARK (Experimental): Parents receive a narrated training program about children's racial biases and read books that are focused on race with their children.
  Interventions: Behavioral: EmBARK
- Popular guidance (Experimental): Parents receive interesting popular press articles about children's racial biases and read books that are focused on race with their children.
  Interventions: Behavioral: Popular guidance
- Practice first (Experimental): Parents practice discussing books about animals with their children first, and then receive a narrated training program about children's racial biases and read books that are focused on race with their children.
  Interventions: Behavioral: Practice first

INTERVENTIONS:
Behavioral: EmBARK — The narrated training teaches parents about children's biases and introduces multiple strategies for addressing children's biases. Families receive children's books to help practice the strategies.
  Arms: EmBARK
Behavioral: Popular guidance — The popular press articles teach parents about children's biases and guide parents about how to talk to children about race. Families receive children's books focused on race to help practice talking about race.
  Arms: Popular guidance
Behavioral: Practice first — Animal books are provided to parents to help them practice talking to their children when reading books. Then, families receive a training program about race as well as children's books about race.
  Arms: Practice first

SUMMARY:
The goal of this clinical trial is to test a parent-led program for reducing children's racial biases in White families. The main question it aims to answer is: With training, can parents effectively address their children's racial biases? Parent will receive training and tools for addressing their children's racial biases. Researchers will study effects on both parents' and children's racial biases.

ELIGIBILITY:
Inclusion Criteria:

* The child is 5.00 to 7.99 years of age
* The child participant and their parent are both non-Hispanic White

Exclusion criteria are:

* Non-proficiency in English on the part of the parent or the child
* The parent is <18 years old
* The child or parent identifies with another racial/ethnic identity in addition to White

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 648 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Likelihood of Child's Racial Bias | Baseline, Post-Test 1 (up to 4 weeks on study), Post-Test 2 (up to 16 weeks on study)
  Total possible range of scores from 1-5. Higher scores mean higher likelihood of bias.
Change in Concern about Children's Racial Bias | Baseline, Post-Test 1 (up to 4 weeks on study), Post-Test 2 (up to 16 weeks on study)
  Total possible range of scores from 1-10. Higher scores indicate more concern.
Change in Concern about Own Child's Bias | Baseline, Post-Test 1 (up to 4 weeks on study), Post-Test 2 (up to 16 weeks on study)
  Total possible range of scores from 1-10. Higher scores indicate more concern.
Change in Motivation to Regulate Children's Bias | Baseline, Post-Test 1 (up to 4 weeks on study), Post-Test 2 (up to 16 weeks on study)
  Total possible range of scores from 1-10. Higher scores mean greater motivation.
Change in Self-Efficacy for Addressing Children's Bias | Baseline, Post-Test 1 (up to 4 weeks on study), Post-Test 2 (up to 16 weeks on study)
  Total possible range of scores from 1-7. Higher scores mean greater self-efficacy.
Change in Intergroup Liking | Baseline, Post-Test 1 (up to 4 weeks on study), Post-Test 2 (up to 16 weeks on study)
  Total possible range of scores is -12 to +12. Higher scores reflect more ingroup liking.
Change in Diversity Preference | Baseline, Post-Test 1 (up to 4 weeks on study), Post-Test 2 (up to 16 weeks on study)
  Total possible range of scores is 0 to 4. Higher scores mean a greater preference for homogeneous groups.
Change in Reactions to Discrimination: Evaluation | Baseline, Post-Test 1 (up to 4 weeks on study), Post-Test 2 (up to 16 weeks on study)
  Total possible range of scores is -6 to +6.
Change in Reactions to Discrimination: Confrontation | Baseline, Post-Test 1 (up to 4 weeks on study), Post-Test 2 (up to 16 weeks on study)
  Participants can score 0 or 1, with the higher score reflecting confrontation.
Change in Predicting Parents' Attitudes | Post-Test 1 (up to 4 weeks on study), Post-Test 2 (up to 16 weeks on study)
  Total possible range of scores is -6 to +6.

CONTACTS AND LOCATIONS:
Locations (1):
- Waisman Center at UW-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data collected during the trial, after de-identification, will be shared. Additionally, the study protocol, statistical analysis plan, informed consent form, and analytic code will be shared. The materials will be shared upon publication of primary outcomes, and will be available indefinitely. They will be shared via an open science platform, namely the Open Science Framework (OSF). Anyone may access the data to verify study outcomes or make additional data discoveries.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The materials will be shared upon publication of primary outcomes, and will be available indefinitely.
Access Criteria: The data will be shared via an open science platform, namely the Open Science Framework (OSF). Anyone may access the data to verify study outcomes or make additional data discoveries.